CLINICAL TRIAL: NCT05295329
Title: Effect of Compound Danshen Dripping Pills on Diabetic Patients With Coronary Microcirculation Disturbance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDDP-202012
Record Dates: First submitted 2022-03-01; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2021-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Take compound salvia miltiorrhiza dropping pills
  Interventions: Drug: Compound Danshen Dropping Pills
- placebo group (Placebo Comparator): Take a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Compound Danshen Dropping Pills — use Compound Danshen Dropping Pills
  Arms: Test group
Drug: Placebo — use placebo
  Arms: placebo group

SUMMARY:
Most patients with diabetes complicated with microvascular circulation disorder have normal coronary angiography but still suffer from chest tightness, chest pain and so on. Early dysfunction of coronary microcirculation is an important reason for it. It is also an important factor leading to poor prognosis of patients with diabetes. For these patients, there are still no drugs to improve microcirculation disorders. Compound Danshen dropping pills have the effects of anti-oxidation, anti-inflammatory, protecting endothelium, inhibiting the formation of atherosclerotic plaque and intimal hyperplasia, reducing oxygen consumption, improving energy metabolism, protecting cardiomyocytes, inhibiting platelet adhesion and aggregation, and improving microcirculation. However, there is a lack of clinical evidence that compound Danshen dripping pills can improve the cardiac microcirculation disturbance in diabetic patients with microangio angina. Therefore, the aim of this study was to observe the effect of Compound Danshen Dripping Pills on coronary microcirculation disturbance in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: 1) age ≥ 18 and ≤ 75, male or female. 2) The microcirculation resistance index (IMR) of the left anterior descending coronary artery was ≥ 25.

  3) the diagnosis of type 2 diabetes or type 2 diabetes has been confirmed. 4) Combined with chest tightness, chest pain, palpitation, shortness of breath and other typical or atypical symptoms of angina pectoris.

  5) Coronary angiography showed no severe epicardial coronary artery stenosis (diameter stenosis rate < 50%).

  6) The patient himself agreed to participate in this study.

Exclusion Criteria:

* Subjects that meet any of the following criteria will be excluded from this study:

  1. Severe cardiac insufficiency (LVEF<40%).
  2. Atrioventricular block and bronchial asthma above II°. (3) Malignant hypertension (SBP≥200 mmHg and/or DBP≥120 mmHg) or severe hypotension (SBP < 90 mmHg).

  4) Acute myocarditis, pericardial disease, valvular heart disease, primary cardiomyopathy, myocardial infarction, severe left ventricular hypertrophy (ventricular wall or septum thickness ≥13mm).

  5) Familial hypercholesterolemia. 6) Multiple arteritis. 7) Heart stenting was performed within 3 months. 8) Coronary artery bypass grafting. 9) History of stroke within six months, history of intracranial diseases (aneurysm, arteriovenous malformation), history of extensive trauma or surgery within six weeks; 10) Active bleeding, anemia of moderate or higher severity, including known thrombocytopenia or leukopenia, severe liver or kidney dysfunction, uncontrolled infection, immune system and connective tissue diseases.

  11) those who are pregnant or lactation, or have the intention to give birth within one year, or take effective contraceptive measures during their childbearing years.

  12) Abnormal liver function (serum ALT level exceeding 3.0 times the upper limit of normal) or abnormal kidney function (eGFR≤30%).

  13) Other respiratory, digestive, blood, infectious, immune, endocrine, neuropsychiatric, tumor and other diseases of clinical significance, which may cause serious risks to patients.

  14) Patients requiring warfarin or NOAC anticoagulation treatment are taking K channel opening agents and Traditional Chinese medicine preparations for promoting blood circulation and removing stasis to improve microcirculation.

  15) Allergic to contrast agent or CDDP; 16) Life expectancy less than one year; 17) Patients who participated in other TCM clinical studies within 12 months prior to inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
IMR improvementcompared with baseline. | 3 months
  Proportion of subjects with ≥ 20% reduction in IMR after 3 months of medication

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Long March Hospital Affiliated to Naval Medical College, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Medical College of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated to Medical College of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Minhang District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Putuo District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided